CLINICAL TRIAL: NCT00184457
Title: Maximal Leg Press Strength Training for Coronary Artery Disease Patients. Training Effect on Serum Testosterone and Work Economy
Brief Title: Maximal Leg Press Strength Training Study for Coronary Artery Disease Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25060100
Record Dates: First submitted 2005-09-15; First posted 2005-09-16 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2011-11

CONDITIONS: Heart Failure; Coronary Artery Disease
Keywords: Cardiac heart failure; Leg press; Maximal strength training; Serum testosterone; Work economy
MeSH Terms: conditions — Heart Failure; Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Strength training intervention

SUMMARY:
Maximal strength training has been shown to increase muscular strength, muscular volume and work economy. An 8 week maximal leg press training regime will be conducted on cardiac heart failure patients to evaluate whether they increase their maximal leg press strength, work economy, serum testosterone and quality of life. The study hypotheses are that:

1. Aerobic work capacity will increase due to increased work economy, without increases in maximal oxygen uptake.
2. Strength training will increase serum testosterone.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed coronary artery disease
* Stable coronary artery disease
* 1.5 mm depression in ST segment during a cycling strain test
* Between 18-70 years of age

Exclusion Criteria:

* Unstable coronary artery disease
* Other limitations to exercise than coronary artery disease
* Participants in other study interventions

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2005-09; Primary Completion 2007-04 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Maximal leg press strength
Work economy
Serum testosterone
Quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Asbjørn Støylen, MD, Study Director — Norwegian University of Science and Technology
Locations (1):
- Norwegian University of Science and Technology, Trondheim, Norway

REFERENCES:
- [Result] Karlsen T, Helgerud J, Stoylen A, Lauritsen N, Hoff J. Maximal strength training restores walking mechanical efficiency in heart patients. Int J Sports Med. 2009 May;30(5):337-42. doi: 10.1055/s-0028-1105946. Epub 2009 Feb 6. PMID 19199203